CLINICAL TRIAL: NCT03919604
Title: Extracorporeal Membrane Oxygenation for Lung Transplantation in Cystic Fibrosis Patients: Predictors and Impact on Outcome
Brief Title: ECMO for Lung Transplantation in Cystic Fibrosis Patients
Acronym: RetroLUTX
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, Chief of Critical Care Unit, Policlinico Hospital
Other Study IDs: 346_2018bis
Record Dates: First submitted 2019-04-11; First posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; lung transplantation; extracorporeal membrane oxygenation
MeSH Terms: conditions — Cystic Fibrosis | interventions — Extracorporeal Membrane Oxygenation; Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECLS group: Patients with CF undergoing LUTX. Need for intraoperative extracorporeal life support
  Interventions: Procedure: Extracorporeal Life Support
- Non-ECLS group: Patients with CF undergoing LUTX. No need for intraoperative extracorporeal life support

INTERVENTIONS:
Procedure: Extracorporeal Life Support — Any extracorporeal blood treatment technique for respiratory and/or cardiac support
  Other Names: Extracorporeal membrane oxygenation; Cardiopulmonary Bypass
  Groups: ECLS group

SUMMARY:
Cystic fibrosis (CF) is the most common genetically inherited disease in the Caucasian population. Bilateral lung transplantation (LUTX) is a viable option for these patients.

Frequently, the surgical operation of LUTX is complicated by hemodynamic instability, intractable hypoxia and respiratory acidosis. For these reasons, Intraoperative extracorporeal life support - ECLS- is required. Data on predictors of use of intraoperative ECLS in CF patients undergoing LUTX is scarce. Aim of this retrospective observational study was 1) to find possible risk factors at the time of enlistment associated with the intraoperative use of ECLS and 2) to compare the outcomes of CF patients treated with ECLS during LUTX or not.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most common genetically inherited disease in the Caucasian population and damages multiple organ systems (i.e., upper and lower respiratory tract, pancreas, liver). Respiratory manifestations include reduction of mucus clearance, chronic pulmonary infections and bronchiectasis, causing progressive respiratory failure that is the primary cause of death in CF patients. Moreover, advanced CF is complicated by pulmonary hypertension, right ventricular hypertrophy and right heart failure. Bilateral lung transplantation (LUTX) is a viable option for these patients, providing a significant survival benefit as compared to no-LuTX.

Frequently, the surgical operation of LUTX is complicated by acute heart failure (due to sequential pulmonary artery cross-clamping and/or hemodynamic instability), severe intractable hypoxia and respiratory acidosis. For these reasons, extracorporeal life support - ECLS - (either in the form of cardiopulmonary bypass -CBP- or extracorporeal membrane oxygenation -ECMO) is frequently required.

To now, literature data on predictors of use of intraoperative ECLS in CF patients undergoing LUTX is scarce. Notably, the use of ECLS during LUTX has been associated with a higher risk of primary graft dysfunction (PGD). Moreover, knowing that a patient has a high risk for the use of ECLS may allow appropriate clinical planning of the procedure with eventual elective ECMO connection.

The investigator's Institution (Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico) is an Italian tertiary referral center for CF and LUTX, as well as for respiratory failure and ECMO support. Aim of this retrospective observational study was 1) to find possible risk factors at the time of enlistment associated with the intraoperative use of ECLS and 2) to compare the outcomes of CF patients treated with ECLS during LUTX or not.

ELIGIBILITY:
Inclusion Criteria:

* CF
* undergoing LUTX

Exclusion Criteria:

* single lung transplantation
* re-transplantation
* missing medical records.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with CF undergoing LUTX at Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico during the study period
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Intraoperative use of blood components | Jan 2013 Dec 2018
  Intraoperative use of: 1) packed red blood cells used (units); 2) fresh frozen plasma (units); 3) pooled platelets (units)
Length of mechanical ventilation | Jan 2013 Dec 2018
  Length of invasive mechanical ventilation (days)
Length of intensive care unit (ICU) stay | Jan 2013 Dec 2018
  Intensive care unit stay (days)
Length of Hospital stay | Jan 2013 Dec 2018
  Length of hospital stay (days)
Primary graft dysfunction | Jan 2013 Dec 2018
  Primary graft dysfunction at 72 hours from re-perfusion of grafts (classes)

SECONDARY OUTCOMES:
Survival | Jan 2013 Dec 2018
  survival at 31st March 2019.

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Grasselli, Study Director — Universita' di Milano
Locations (1):
- Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided